CLINICAL TRIAL: NCT06792409
Title: Motiva Mia® Pilot Study to Evaluate the Safety and Initial Effectiveness of the Procedure and System Devices, Including Motiva Implants® Ergonomix2 Diamond® in Subjects Undergoing Primary Breast Augmentation Procedures
Brief Title: Mia® Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Establishment Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLINP-001007 CR
Record Dates: First submitted 2024-12-11; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Augmentation
Keywords: Mia; Breast; augmentation; Minimally invasive; Transaxillar; Transaxillary; Motiva; Injector; Balloon; Inflatable Balloon; Ergonomix2; Implants; Dissector; Implant; Silicone; Diamond

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minimally Invasive breast augmentation (Experimental): Minimally invasive breast augmentation procedure with a trans-axillary approach.
  Interventions: Device: Minimally invasive breast augmentation procedure with a trans-axillary approach.

INTERVENTIONS:
Device: Minimally invasive breast augmentation procedure with a trans-axillary approach. — Minimally invasive breast augmentation procedure with a transaxillary approach using Motiva Ergonomix2 Diamond®, Motiva Injector® and Motiva® Inflatable Balloon.
  Other Names: Inflatable Balloon; Injector; Ergonomix breast implants

SUMMARY:
This study will follow 100 women over 36 months (3 years) to evaluate how safe and effective a minimally invasive breast augmentation procedure is. The women will have their first breast augmentation surgery using Motiva® Ergonomix2 Diamond® implants, Motiva Injector® and Motiva® Inflatable Balloon.

DETAILED DESCRIPTION:
This is a prospective follow-up, 36-month, open, interventional study to confirm the safety and effectiveness of the procedure and system devices, including Motiva® Ergonomix2 Diamond® implants in women subjected to primary breast augmentation.

This study will enroll 100 women who will undergo a minimally invasive breast augmentation procedure with Ergonomix2 Diamond® using Motiva Injector® MIA and the Motiva MIA® inflatable balloon. The study duration will be 36 months and a six-month enrollment window was planned.

Recruitment will take place after enrollment and before any clinical research procedures, a participant will sign and date the Informed Consent Form. This will be considered the intent-to-treat (ITT) population. Since there will be a subset of women who will provide their consent to participate but will not undergo the procedure (i.e., due to a screening failure or consent withdrawal before the surgery, the analysis population for this study will be the full analysis set ("treated population") which will be made up by women that have received the implant(s) and that have at least one postop evaluation.

A Magnetic Resonance Imaging (MRI) substudy will be performed to determine the rate of silent rupture (no signs or symptoms) both extra- and intracapsular, and to identify displacement and/or gel fracture. MRI scans in this study will be performed on participants who are 18 to 21 months post-op. However, any study participant, whether or not participating in this sub study, who presents with signs or symptoms suggestive of a rupture, will be referred for MRI evaluation at any time during the study. Information obtained from the MRI study will be collected on the MRI Case Report Form by the investigator.

The proposed sample size of 33 participants in the MRI substudy, considered to be the industry standard, one third of the total sample participating in the Motiva MIA® study, and who consent to participate in this substudy.

ELIGIBILITY:
Inclusion Criteria:

* Genetic females, ≥ 18 years.
* AA to C cup size, evaluated according to Triumph international guidelines.
* Participants with Class I and II risk according to the American Society of Anesthesiologists (ASA)
* Participants seeking a primary breast augmentation to increase the size of their breasts by one cup size.
* Body Mass Index between 18.5 and 24.9 (normal weight).
* Adequate tissue for covering the implant(s).
* Willingness to follow all study requirements and attending all necessary follow-up visits.
* Agreement to return the device to the sponsor in case it is explanted

Exclusion Criteria:

* Current costal lesions.
* Breast ptosis or poor skin quality.
* Inadequate tissue (for example, radiation damage, ulcers, compromised vascularity, history of inadequate wound scaring).
* History of abscesses or infections in the breast area.
* Currently pregnant or breastfeeding, or pregnancy or breastfeeding to term in the six months prior to recruitment.
* History of silicone sensitivity.
* Use of any medications that interfere with coagulation or that may imply a high risk and/or significant post-surgical complication.
* Any medical condition, such as low weight or obesity according to the inclusion criteria, diabetes, autoimmune disease, chronic lung disease or serious cardiovascular disease that may result in an excessively high surgical risk and/or important post-surgical complications.
* Any condition that precludes the use of magnetic resonance imaging (MRI), including implanted metal devices, claustrophobia or other conditions that preclude MRI exploration.
* Any history of psychological characteristics that are not realistic or reasonable, considering the risks involved with the surgical procedure.
* Use of any medications that, according to the investigator, may imply a higher risk of complications or interference with wound healing ability, such as corticosteroids or anticoagulants (i.e., concomitant warfarin therapy).
* Current participation on studies for investigation devices or pharmaceutical products.
* Participants not residing in Costa Rica, which precludes their attendance to follow-up visits.
* Sponsor (or any of its subsidiaries) employees, study investigator or any person helping to conduct the study; direct (family) relationship with any sponsor (or any of its subsidiaries) or investigator employees.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetic females, ≥ 18 years.
Enrollment: 100 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Safety | From minimally invasive procedure through study completion, an average of 3 years.
  Cumulative incidence (number of cases) of adverse events during surgery and the follow-up period, severity and duration of all complications (rate of adverse events related to the procedure / adverse events related to the device).
Effectiveness | From minimally invasive procedure through study completion, an average of 3 years.
  Effectiveness will be measured as satisfactory on all breast augmentation procedures using Mia® devices if no device failures have occurred.

SECONDARY OUTCOMES:
Patient satisfaction | From week 1 post-procedure to the end of the follow-up period
  Percentage of participants in the BREAST-Q© augmentation model according to the scale.
Patient satisfaction | From week 1 post-procedure to the end of the follow-up period
  Central trend (mean) of participants in the BREAST-Q© augmentation model according to the scale.
Patient satisfaction | From week 1 post-procedure to the end of the follow-up period
  Variability (standard deviation) of participants in the BREAST-Q© augmentation model according to the scale.
Surgeon satisfaction | During minimally invasive procedure
  Surgeon satisfaction with the results of the minimally invasive procedure using the satisfaction 5-item Likert scale, named Global Aesthetic Improvement Scale (GAIS).

OTHER OUTCOMES:
Device Malfuctioning | During minimally invasive procedure
  Finalizing the expected placement of the breast implant without the device malfunctioning.
Use of conventional surgical techniques | During minimally invasive procedure
  Finalizing the expected placement of the breast implant without the need for correcting or adjusting using conventional surgical techniques.
Surgical pocket | During minimally invasive procedure
  Performing a surgical pocket dissection procedure to adequately place the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Europeo de Cirugía, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: Yes
Once the study is complete, the sponsor will analyze the data collected by the principal investigator and will conduct a scientific publication with all parties involved to unveil the study results.